CLINICAL TRIAL: NCT02637908
Title: Head Start Parenting
Brief Title: Mindfulness Training for Head Start Parents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2014-1287
Record Dates: First submitted 2015-09-03; First posted 2015-12-22 (Estimated); Last update posted 2016-08-10 (Estimated); Status verified 2016-08

CONDITIONS: Stress, Physiological
Keywords: Mindfulness; Parents; Families

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mindfulness training (Experimental): The mindfulness training (experimental condition) will receive 6-weeks of mindfulness training for parents provided in a group setting.
  Interventions: Behavioral: Mindfulness training
- Wait-list control (No Intervention): The wait-list control group will receive no intervention during the course of the study. The control group will be offered training following the completion of the study.

INTERVENTIONS:
Behavioral: Mindfulness training — 6-weeks of group-based mindfulness training for parents
  Arms: Mindfulness training

SUMMARY:
A training module has been developed for parents to effectively address stressors and demands of parenting and promote positive and supportive parent-child interactions. The purpose of this study is to implement the parent training program and evaluate the effectiveness of the program. Depending on the results, investigators expect core aspects of this module to be adaptable and modified or extended for parents of older children in the future to meet the needs of families across the stages of childhood development.

DETAILED DESCRIPTION:
Parents of children enrolled in the Head Start program will be recruited to take part in a training module to learn and practice mindfulness techniques. Recruited participants will be randomly assigned to an intervention group or a wait-list control group. Parents in the intervention group will attend the training, which involves 6 weekly, group sessions. Data will be collected from both the intervention and wait-list control groups 1-3 weeks prior to the intervention period and 1-3 weeks following the end of the intervention period. This data will be collected through self-report questionnaires, in-home observations, hair sample from parents, an activity tracker for parents, and records on developmental assessments and attendance of the target child from Head Start. The wait-list control group will be offered a training after measures are completed. Intervention group participants may be invited to take part in focus groups after the training is complete. At these focus groups, they will engage in a discussion of their experiences and opinions about the class. Some participants may be invited to individual interviews to share their experiences and aid further revision of the program.

ELIGIBILITY:
Inclusion Criteria:

* Parents of children ages 0 - 5 who are enrolled in Head Start

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2015-09; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Change in Parent Relationship Questionnaire 2-5 (PRQ2-5) scores (Kamphaus & Reynolds, 2006) | 1-3 weeks prior to intervention; 10 - 13 weeks after baseline (1-3 weeks post-intervention)
  The PRQ2-5 will be completed by the parent participant prior to the intervention period and directly following the end of the intervention period in order to assess any change in the parent-child relationship.
Change in HOME Infant / Toddler / Early Childhood Record Form scores (Totsika & Sylva, 2004) | 1-3 weeks prior to intervention; 10 - 13 weeks after baseline (1-3 weeks post-intervention)
  Observations of parents and children will be completed in parents' homes prior to the intervention and directly following the intervention period. Observations will involve completion of the HOME Record Form by trained observers. The observations completed at each time point will be used to assess change in the home environment of the child.
Change in Symptom Checklist 90 Revised (SCL-90 R) scores (Derogatis, 1994) | 1-3 weeks prior to intervention; 10 - 13 weeks after baseline (1-3 weeks post-intervention)
  Parents will complete a self-report questionnaire assessing their own psychological symptoms prior to the intervention period and directly following the end of the intervention. Scores acquired at each time point will be used to assess change in the parent participant's psychological symptoms.
Change in Psychological Well-Being Scales scores (Ryff & Keyes, 1995) | 1-3 weeks prior to intervention, 10 - 13 weeks after baseline (1-3 weeks post-intervention)
  Parents will complete a self-report questionnaire assessing their level of psychological well-being prior to the intervention period and directly following the end of the intervention. Scores acquired at each time point will be used to assess change in the parent participant's psychological well-being.

SECONDARY OUTCOMES:
Change in physical activities and characteristics measured using FitBit Activity Tracker (Bai et al., 2015) | Worn for 5 days at 1-3 weeks prior to intervention; worn for 5 days at 10 - 13 weeks after baseline (1-3 weeks post-intervention)
  Data will be collected on the parent's physical activity, including steps, sleep and heart rate, using a FitBit Activity Tracker device. The data collected at each time point will be used to assess change in the parent participant's physical activity.
Change in Prescription medication use | 1-3 weeks prior to intervention; 10 - 13 weeks after baseline (1-3 weeks post-intervention)
  Parents' self-report of their prescription medication use will be collected prior to the intervention and directly following the end of the intervention period. Information collected at each time point will be used to assess any change in the parent participant's prescription medication use.
Adverse Childhood Experiences (Edwards, et al., 2003) | 1-3 weeks prior to intervention
  The Adverse Childhood Experiences questionnaire will be completed by parents to assess the parents' childhood experiences prior to the intervention.
Family Instability Questionnaire (Ackerman et al., 1999) | 1-3 weeks prior to intervention
  Parents will complete a self-report questionnaire assessing events related to family instability that may have taken place prior to the intervention period.
Family Instability Questionnaire (Ackerman et al., 1999) | 10 - 13 weeks after baseline (1-3 weeks post-intervention)
  Parents will complete a self-report questionnaire assessing events related to family instability that may have taken place during the time of the intervention period.
Change in Pittsburgh Sleep Quality Index scores (Buysse et al., 1989) | 1-3 weeks prior to intervention; 10 - 13 weeks after baseline (1-3 weeks post-intervention)
  Parents will complete a self-report questionnaire assessing their own sleep quality prior to the intervention period and directly following the end of the intervention period. Data collected at each time point will be used to assess changes in the parent participant's sleep quality.
Change in Five Facet Mindfulness Questionnaire scores (Baer et al., 2008) | 1-3 weeks prior to intervention; 10 - 13 weeks after baseline (1-3 weeks post-intervention)
  Parents will complete a self-report questionnaire assessing their level of mindfulness prior to the intervention period and directly following the end of the intervention. Scored collected at each time point will be used to assess changes in the parent's level of mindfulness.
Hair cortisol (Russell et al., 2012) | 10 - 13 weeks after baseline (1-3 weeks post-intervention)
  Cortisol will be assessed in the hair of consenting parents directly following the end of the intervention period.
Change in Behavior Assessment System for Children scores (Reynolds & Kamphaus, 2004) | 1-3 weeks prior to intervention; 10 - 13 weeks after baseline (1-3 weeks post-intervention)
  Parents will complete a questionnaire concerning observed behaviors of their child prior to the intervention period and directly following the end of the intervention. Scores collected at each time point will be used to assess any change in the parent participant's perception of the target child's behavior.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Flook, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- Dane County Parent Council Inc, Madison, Wisconsin, United States

REFERENCES:
- [Background] Reynolds, C. R., & Kamphaus, R. W. (2004). BASC-2. Behavioral Assessment System for Children (2nd ed.). Circle Pines, MN: AGS.
- [Background] Kamphaus, R. W., & Reynolds, C. R. (2006). Parenting relationship questionnaire (PRQ). Bloomington, MN: Pearson Assessments.
- [Background] Bai Y, Welk GJ, Nam YH, Lee JA, Lee JM, Kim Y, Meier NF, Dixon PM. Comparison of Consumer and Research Monitors under Semistructured Settings. Med Sci Sports Exerc. 2016 Jan;48(1):151-8. doi: 10.1249/MSS.0000000000000727. PMID 26154336
- [Background] Totsika V, Sylva K. The Home Observation for Measurement of the Environment Revisited. Child Adolesc Ment Health. 2004 Feb;9(1):25-35. doi: 10.1046/j.1475-357X.2003.00073.x. PMID 32797621
- [Background] Ackerman BP, Kogos J, Youngstrom E, Schoff K, Izard C. Family instability and the problem behaviors of children from economically disadvantaged families. Dev Psychol. 1999 Jan;35(1):258-68. doi: 10.1037//0012-1649.35.1.258. PMID 9923480
- [Background] Derogatis, L. R. (1994). SCL-90-R Symptom Checklist-90-R administration, scoring and procedures manual. Minneapolis, MN: National Computer Systems.
- [Background] Edwards VJ, Holden GW, Felitti VJ, Anda RF. Relationship between multiple forms of childhood maltreatment and adult mental health in community respondents: results from the adverse childhood experiences study. Am J Psychiatry. 2003 Aug;160(8):1453-60. doi: 10.1176/appi.ajp.160.8.1453. PMID 12900308
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Background] Russell E, Koren G, Rieder M, Van Uum S. Hair cortisol as a biological marker of chronic stress: current status, future directions and unanswered questions. Psychoneuroendocrinology. 2012 May;37(5):589-601. doi: 10.1016/j.psyneuen.2011.09.009. Epub 2011 Oct 4. PMID 21974976
- [Background] Baer RA, Smith GT, Lykins E, Button D, Krietemeyer J, Sauer S, Walsh E, Duggan D, Williams JM. Construct validity of the five facet mindfulness questionnaire in meditating and nonmeditating samples. Assessment. 2008 Sep;15(3):329-42. doi: 10.1177/1073191107313003. Epub 2008 Feb 29. PMID 18310597
- [Background] Ryff CD, Keyes CL. The structure of psychological well-being revisited. J Pers Soc Psychol. 1995 Oct;69(4):719-27. doi: 10.1037//0022-3514.69.4.719. PMID 7473027